CLINICAL TRIAL: NCT05057195
Title: Wide Excision of Soft Tissue Sarcomas in Combination With Interstitial Radiation Therapy in Patients With Soft Tissue Sarcomas of the Upper and Lower Extremities Compared With Postoperative Radiation Therapy
Brief Title: Wide Excision of Soft Tissue Sarcomas in Combination With Interstitial Radiation Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Blokhin's Russian Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SARCBT-2021-7-11
Record Dates: First submitted 2021-09-07; First posted 2021-09-27 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Sarcoma; Soft Tissue Sarcoma
Keywords: Sarcoma; Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interstitial radiation therapy (Experimental): Duration: 11 days
  Interventions: Radiation: Interstitial radiation therapy
- Postoperative external beam therapy, on the bed of the removed tumor (Active Comparator): Duration: 4 weeks
  Interventions: Radiation: Postoperative external beam therapy

INTERVENTIONS:
Radiation: Interstitial radiation therapy — From 30 to 50 Gy,
  Arms: Interstitial radiation therapy
Radiation: Postoperative external beam therapy — 50 Gy and locally on the tumor bed up to 10-26 Gy, depending on the status of the resection margin
  Arms: Postoperative external beam therapy, on the bed of the removed tumor

SUMMARY:
Intraoperatively, in the bed of the removed tumor, a surgical mesh is sutured onto which the intrastats are fixed. On days 2-3, topometric preparation is carried out, the choice of the amount of irradiation, the calculation of the program. On the 4-5th day after the operation, a course of intra-tissue radiation therapy begins in a single dose of 3 to 5 Gy in 10 fractions 2 times a day with an interval between fractions of 6 hours, the planned total dose is from 30 to 50 Gy. (from 40 to 70 IGy). Follow-up examination after 4 weeks and then every 3 months for 24 months

DETAILED DESCRIPTION:
1 day before the operation, taking blood tests: general blood test with counting the leukocyte formula and the number of platelets; biochemical blood test with the determination of indicators of liver and kidney function (including electrolytes); coagulogram; performing surgical treatment with urgent histological examination of the edge of the tumor; intraoperatively, in the bed of the removed tumor, a surgical mesh is sutured onto which the intrastats are fixed with the fixation of the outlet ends on the skin with the help of buttons. 1 day after the operation, taking blood tests: a general blood test with the calculation of the leukocyte formula and the number of platelets; biochemical blood test with the determination of indicators of liver and kidney function (including electrolytes); coagulogram.

On the 2-3rd day after the surgical treatment, topometric preparation, the choice of the amount of radiation, and the calculation of the program are carried out. On the 4-5th day after the operation, a course of interstitial radiation therapy begins in a single dose of 3 to 5 Gy in 10 fractions 2 times a day with an interval between fractions of 6 hours, the planned total dose is from 30 to 50 Gy, which is equivalent to 40 to 70 IGy (isogrey). On the 6th day, removal of intrastats, on the 7th day after the operation, ultrasound of the wound and n / c vessels; assessment of the nature of wound healing. On the 10th day, discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* C49.1 Malignant neoplasm of the connective and soft tissues of the upper limb, including the shoulder girdle
* C49.2 Malignant neoplasm of the connective and soft tissues of the lower limb, including the hip region
* Tumor size 7 cm or less
* For malignant tumors: Grade 2-3
* Locally advanced soft tissue sarcomas
* Absence of regional metastases
* Tumor recurrence

Exclusion Criteria:

* Children, women during pregnancy, childbirth, women during breastfeeding.
* Military personnel, with the exception of contract military personnel.
* Persons with mental disorders.
* Persons detained, taken into custody, serving a sentence in the form of restriction of freedom, arrest, imprisonment or administrative arrest.
* The age of patients is under 18 years old
* Histologically confirmed diagnosis of GIST, Kaposi's sarcoma, alveolar, clear cell sarcoma, chondrosarcoma, paraossal osteosarcoma
* Inoperable tumor
* A tumor with decay or with the threat of decay
* The presence of damage to the skin in the affected area
* The presence of a second malignant tumor
* Having an active or chronic fungal / bacterial / viral infection
* Uncontrolled chronic diseases of the liver, kidneys in the acute stage
* Superficial tumor (within the skin)
* The use of a reconstructive plastic component using a displaced musculocutaneous flap
* The use of vascular prosthetics
* The removed tumor bed is more than 7 cm
* The presence of a tumor growing into the bone
* The presence of blood vessels and nerves in the removed tumor bed
* Presence of metastases
* Surgical intervention using transplanted skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 24 months
  Time after treatment during which no sign of cancer is found

SECONDARY OUTCOMES:
Comparison of hospitalization rate | 30 days
  Time after surgery till the end of hospitalization
Comparison of safety assessment | 24 months
  Adverse Event Assessment and Serious Adverse Event Assessment according to CTCAE 5.0
Comparison of performance status according Karnofsky scale | 24 months
  Improvement on the Karnofsky scale by 10-30 points
Comparison of pain relief according Visual Analogue Scale | 24 months
  Improvement on the Visual Analogue Scale by 3-5 points
Comparison of pain relief according Whatkins scale | 24 months
  Improvement on the Whatkins scale by 1-2 points

CONTACTS AND LOCATIONS:
Overall Officials: Aslan Valiev, PhD, Principal Investigator — N.N. Blokhin NMRCO
Locations (1):
- Federal State Budgetary Institution "N.N. Blokhin National Medical Research Center of Oncology" оf the Ministry of Health of the Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: official site — https://www.ronc.ru/about/struktura/niiko/ooo/hn1/
- See also: russian surcoma group site — https://sarcomarus.ru/